CLINICAL TRIAL: NCT00334204
Title: Does An Abnormal PFA 100 Predict Bleeding After Renal Biopsy?
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: run out of independent funding
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Tibor Fulop, Associate Professor of Medicine, University of Mississippi Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2004-0092
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Results first posted 2013-08-01 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-06

CONDITIONS: Kidney Failure, Acute; Kidney Failure, Chronic; Blood Platelet Disorders; Hemorrhage
Keywords: Platelet Function Analyser-100 (PFA-100); renal failure; kidney biopsy; bleeding; hematoma
MeSH Terms: conditions — Acute Kidney Injury; Kidney Failure, Chronic; Blood Platelet Disorders; Hemorrhage; Renal Insufficiency; Hematoma | interventions — Platelet Function Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Measure Platelet Function Analyser -100 (PFA-100) (Other): measuring Platelet Function Analyser (PFA)-100 test (an in vitro platelet function test, in addition to the rest of the routine/uusal clinical care)
  Interventions: Device: measuring Platelet Function Analyser-100 (PFA-100) platelet function before kidney biopsy

INTERVENTIONS:
Device: measuring Platelet Function Analyser-100 (PFA-100) platelet function before kidney biopsy — measuring Platelet Function Analyser (PFA) -100 platelet function before kidney biopsy
  Other Names: in vitro platelet tests; platelet closure time; platelet function

SUMMARY:
The kidneys are highly vascular organs and any trauma or surgery poses risk of severe bleeding. Platelet function is an integral part of the blood clotting during the initial, so-called vascular phase. So far no universally accepted, easy test has been available to measure platelet functions. Renal failure is a condition generally associated with bleeding due to platelet dysfunctions. This study is exploring the utility of a novel platelet function test, called Platelet Function Analyser-100 to predict bleed after percutaneous kidney biopsy. Platelet Function Analyser-100 will be measure before kidney biopsy along with routine blood tests. Subjects will undergo renal ultrasound before and after renal biopsy to verify post-biopsy bleeding events.

DETAILED DESCRIPTION:
Many patients with advanced chronic kidney disease have a predisposition to bleed. This predisposition becomes problematic when they have to undergo an invasive procedure such as a renal biopsy. There are multiple factors that play a role in the predisposition to bleed. These factors all cause abnormal platelet function. Historically there are several tests that have been used to assess the bleeding tendency of patients with renal disease. The most extensively studied of these is the bleeding time. Ideally this is not the best test because it is difficult to reproduce, insensitive, operator dependent and time consuming. Recognizing the limitation of the bleeding time, the Platelet Function Analyser-100 (PFA-100) was developed. This test attempts to mimic the way a clot normally forms in the body.

The purpose of this study is to determine whether an abnormal Platelet Function Analyser-100, a test which determines platelet function, is an accurate predictor of bleeding in those with chronic kidney disease.

All patients admitted for renal biopsy will be offered enrollment in this study. Initial data to include the following will be obtained: age, sex, weight, serum creatinine, activated Prothrombin Time/activated Partial Thromboplastin Time, Complete Blood Count and Platelet Function Analyser-100 closure times. Participants will then be placed in groups (cohorts) based on their calculated Glomerular Filtration Rate and if less than 30 cc/min, Desmopressin [Brand Name: DDAVP] (a drug which appears to improve platelet function) will be given. Post-procedure, participants will be monitored for bleeding by obtaining a Complete Blood Count (CBC) 4 hours and approximately 16 hours post-procedure and monitoring urine for blood. The pre- and post-procedure hematocrit and a post biopsy renal ultrasound will be used to determine whether an abnormal Platelet Function Analyser-100 closure time was predictive of a decrease in hematocrit

There are no additional risks of participation in this study. This study would only involve obtaining additional blood but it would be obtained with blood that would otherwise be obtained prior to renal biopsy. There is no direct benefit from this study to enrolled participants. Besides the Platelet Function Analyser-100 blood test, the patients undergoing renal biopsies will undergo the procedure and post-procedure monitoring per standard of care for renal biopsy at this institution.

Inclusion criteria:

Will offer enrollment to essentially all patients undergoing standard percutaneous renal biopsy here at the University Medical Center. These are:

age 18-80, Body Mass Index>35, Modification of Diet in Renal Diseases (DMDRD)formula-based calculated Glomerualar Filtration Rate (GFR)>10cc/minute, Hematocrit >25, platelet count >100, normal aPT/aPTT,

Exclusion criteria:

essentially the contraindications to a standard percutaneous renal biopsy) known bleeding disorder, history of prior bleeding with procedure or known ongoing bleeding at the time of the procedure, Hematocrit <25, Platelet count <100, abnormal activated Prothrombin Time (aPT)/activated Partial Thromboplastin Time (aPTT) pre biopsy, small kidney(s) < 8.0 cm, multiple bilateral renal cyst or masses, hydronephrosis, active urinary tract infection, recent nonsteroidal anti-inflammatory drug use.

Risk:

The Platelet Function Analyser 100 will require an additional 5-10cc of blood to be drawn. No additional sticks will be done since generally prior to biopsy the patients will have Complete Blood Count, aPT/aPTT and chemistries drawn.

Possible benefits to patients:

There will likely be no benefit for the individual patient. The Platelet Function Analyser 100 is a relatively new test for determining platelet dysfunction and there have been limited studies in dialysis patients. However to date, there have been no studies in those with chronic kidney disease. If a correlation is found between an abnormal Platelet Function Analyser and bleeding instead of giving all patients with compromised Glomerular Filtration Rate, desmopressin, only those with abnormal Platelet Function Analyser would be given desmopressin. In essence, this would decrease the patient incurred expenses of hospitalization. This test may also point out those patients who are high risk for bleed post renal biopsy and may ultimately alter length of in hospital monitoring of patients post biopsy.

Other benefit of this test is that it is a noninvasive, rapid and does not require specialized training to perform the test.

Alternatives:

In lieu of checking Platelet Function Analyser 100, a bleeding time could be done but it has been demonstrated in multiple studies to poorly correlate with bleeding. The results for bleeding time often vary because it is a difficult test to reproduce. Currently, there is no standard, or acceptable, pre-renal biopsy platelet function test done at this Institution.

Consent process:

The patient who will be enrolled in this study have already agreed to undergo a renal biopsy which will be the reason for their hospital admission. They will be allowed to discuss with family members via phone or if they are present at the hospital but it will not be feasible for patients to be allowed to take the consent home and defer biopsy for discussion.

The investigator will have a discussion about the Platelet Function Analyser 100 with all prospective participants prior to renal biopsy being performed. The discussion will include the risks and benefits of having the test performed. The patients will be allowed to ask questions. If consent is given then the Platelet Function Analyser-100 will be drawn.

Cost:

There will be no significant increase in cost. The reagent used to do the test is being donated and the Department of Pathology is willing to do the test without any additional charge to the patient.

Compensation to participants: none.

Data preservation and analysis:

The data obtained during this study will only be available to the Principal investigator and immediate study personnel.

The data will be kept by the Principal investigator in a secured location indefinitely.

The results of the Platelet Function Analyser testings will be in the medical record with the result of the other labs obtained during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

Will offer enrollment to essentially all patients undergoing standard percutaneous renal biopsy here at the University Medical Center. These are:

age 18-80, Body Mass Index (BMI) <35, Modification of Diet in Renal Diseases (MDRD) calculated Glomerular Filtration Rate (GFR) >10 cc/minute/1.73 m2, Hematocrit >25, platelet count >100,000/mm3, normal activated Prothrombin Time (aPT)/activated Partial Thromboplastin Time (aPTT).

Exclusion Criteria:

(essentially the contraindications to a standard percutaneous renal biopsy) known bleeding disorder, history of prior bleeding with procedure or known ongoing bleeding at the time of the procedure, Hematocrit <25, Platelet count <100, abnormal aPT/aPTT pre biopsy, small kidney(s) < 8.0 cm multiple bilateral renal cyst or masses, hydronephrosis, active urinary tract infection, recent nonsteroidal anti-inflammatory drug use.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2004-08; Primary Completion 2008-05 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibor Fulop, Principal Investigator — University of Mississippi Medical Center, Nephrology Division
Locations (1):
- University of Mississipppi Medical Center, Adult Hospital, Jackson, Mississippi, United States

REFERENCES:
- [Derived] Islam N, Fulop T, Zsom L, Miller E, Mire CD, Lebrun CJ, Schmidt DW. Do platelet function analyzer-100 testing results correlate with bleeding events after percutaneous renal biopsy? Clin Nephrol. 2010 Mar;73(3):229-37. doi: 10.5414/cnp73229. PMID 20178723

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 58 parcicipant recruited, 2 excluded due to missing data from analysis
Groups:
- Measure PFA-100: measuring PFA-100 test (an in vitro platelet function test, in addition to the rest of the routine/uusal clinical care)
Period: Overall Study
Arm/Group | Measure PFA-100
Started | 58
Completed | 56
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Measure PFA-100
Number analyzed (Participants) | 56
Age Continuous [Mean (Standard Deviation); unit: years] | 43.68 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Bleeding After Kidney Biopsy on Renal Ultrasound 12 Hours After Biopsy
Time Frame: 12 hours
Measure: Number; unit: participants with hematoma
Arm/Group | Measure PFA-100
Number analyzed (Participants) | 56
participants with hematoma | 11

2. Primary Outcome: Hemoglobin/Hematocrit After Biopsy
Time Frame: 12 hours
Measure: Number; unit: participants with hematuria
Groups:
- Measure Platelet Function Analyser-100 (PFA-100): measuring PFA-100 test (an in vitro platelet function test, in addition to the rest of the routine/uusal clinical care)
Arm/Group | Measure Platelet Function Analyser-100 (PFA-100)
Number analyzed (Participants) | 56
participants with hematuria | 5

3. Primary Outcome: Need for Blood Transfusion
Time Frame: 12
Measure: Number; unit: participants requiring PRBC Transfusion
Arm/Group | Measure Platelet Function Analyser-100 (PFA-100)
Number analyzed (Participants) | 56
participants requiring PRBC Transfusion | 4

ADVERSE EVENTS:
Arm/Group | Measure PFA-100
Serious Adverse Events (participants affected / at risk) | 0/56
Other Adverse Events (participants affected / at risk) | 0/56

LIMITATIONS AND CAVEATS:
Early termination leading to lesser-than-planned numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No